CLINICAL TRIAL: NCT03069157
Title: Evaluation of the Effect of Lung Recruitment and Positive End- Expiratory Pressure (PEEP) on Anesthesia Induced Atelectasis Using Lung Ultrasound in Children Undergoing Major Abdominal Surgery.
Brief Title: Evaluation of the Effect of Lung Recruitment and Positive End- Expiratory Pressure (PEEP) on Anesthesia Induced Atelectasis Using Lung Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Director, Anesthesia and surgical icu, Principal Investigator, Assistant lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-33-2016
Record Dates: First submitted 2017-02-10; First posted 2017-03-03 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia Induced Atelectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer generated numbers and concealed by serially numbered,opague and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelopes will be opened by the nurse, the card inside will determine the patient group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without lung recruitment maneuver (No Intervention): patient ventilation will be maintained After induction of anesthesia all patients will be ventilated using pressure controlled mode targeting tidal volume 6-8 ml/kg with inspiratory to expiratory ( I: E) ratio 1:1.5 without recruitment but with PEEP 5cm H2O.
- recruitment group (Active Comparator): lung recruitment manoeuvre will be performed in patients using continuous positive airway pressure( CPAP) (30) cm H2O for (40) seconds after induction of anesthesia then patient will be converted to pressure controlled mode again with PEEP 5 cm H2O.
  Interventions: Procedure: lung recruitment maneuver

INTERVENTIONS:
Procedure: lung recruitment maneuver — lung recruitment manoeuvre will be performed in patients using continuous positive airway pressure( CPAP) (30) cm H2O for (40) seconds after induction of anesthesia then patient will be converted to pressure controlled mode again with PEEP 5 cm H2O
  Arms: recruitment group

SUMMARY:
Atelectasis is a side effect of general anesthesia which can be found in all types of interventions and patients of all ages.1-3 The reported incidence of anesthesia- induced atelectasis in children varies, ranging from 12 to 42% in sedated and nonintubated patients 5, 6 and from 68 to 100% in children with general anesthesia with tracheal intubation or laryngeal mask.

The aim of this work is to evaluate the effect of lung recruitment on anesthesia induced atelectasis using intraoperative lung ultrasound.

Objectives

* To determine the effect of recruitment on anesthesia induced atelectasis using lung ultrasound.
* To Estimate the change of Pao2 with anesthesia induced lung atelectasis.
* To Estimate the change of Pao2 with lung recruitment.
* To evaluate the feasibility of use of lung ultrasound as a tool to guide optimum lung recruitment.

DETAILED DESCRIPTION:
This a randomized control trial is designed to include 40 children aged from one to four years presented for major abdominal surgery.

Forty patients meeting the inclusion criteria will be randomly assigned into to two equal groups:

Group C (n= 20): Without recruitment maneuver (control group)

Group REC (n= 20): recruitment group

All children will be premedicated with oral midazolam 0.5mg/kg half hour before procedure and atropine at a dose of 0.01-0.02 mg/kg( IM). Continuous electrocardiogram (ECG) , pulse oximetry, non-invasive arterial blood pressure, and temperature monitoring will be applied and all patients will be induced with inhalational anesthetic using Sevoflurane+ oxygen(O2) with mac 2%. After deepening of the anesthesia, intravenous (I.V.) line will be inserted and fentanyl 2μg/kg, muscle relaxant will be given in the form of atracurium 0.5mg/kg and patients will be intubated by appropriate size of endotracheal tube.

After induction of anesthesia all patients will be ventilated using pressure controlled mode targeting tidal volume 6-8 ml/kg with inspiratory to expiratory ( I: E) ratio 1:1.5, and Fio2 1, baseline arterial blood gas will be withdrawn. Patients will be divided into two groups. Group (REC) recruitment group; in this group, lung recruitment manoeuvre will be performed in patients using continuous positive airway pressure( CPAP) (30) cm H2O for (40) seconds after induction of anesthesia then patient will be converted to pressure controlled mode again with PEEP 5 cm H2O22,23. In next assessment time, if still there are atelectatic areas recruitment will be repeated and patient will be maintained at PEEP 10 cm H2O till the end of surgery. In group (C) non recruitment group, patient ventilation will be maintained on aforementioned tidal volume without recruitment but with PEEP 5cm H2O.

Lung ultrasound (LUS) LUS will be performed with the portable echograph MicroMax (SonoSite, M-turbo) using a linear probe of 3 to 6 MHz. Each hemithorax will be divided into six sections using three longitudinal lines (parasternal, anterior, and posterior axillary) and two axial lines, one above the diaphragm and another one 1 cm above the nipples.

As LUS provides regional information, we will repeat the following examination sequence in each hemithorax and in all patients: (1) anterior, (2) lateral, and (3) posterior regions starting from the diaphragm (caudal lung) and moving toward the apex (cranial lung).13,14 Each hemithorax will be assessed using the two-dimensional classical view placing the probe parallel to the ribs .24 (fig. 1).The LUS of a normal lung shows a lung sliding (caused by the respiratory movement of the visceral pleura relative to the fixed parietal pleura) and A lines (repetitive horizontal reverberation artifacts generated by air within the lungs separated by regular intervals, the distances of which being equal that between the skin and the pleural line.

Patients demographic data will be collected; age, gender, weight, height, type of surgery and duration of surgery.

Lung ultrasound examinations will be performed at different time-points immediately before induction of anesthesia, 5, 15 minutes following induction of general anesthesia, before extubation and after extubation at recovery room to detect and monitor atelectasis. Arterial blood samples will be collected simultaneously to measure Pao2.

Atelectasis will be assessed by ultrasound using lung aeration score applied for each region. Lung score is four points (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation) so, applying score for 12 regions bilateral will result in maximum score 36 and lowest score 0.

The sum of surface area of atelectatic regions and the number of recruitment attempts to recruit atelectatic areas will be recorded.

Other data as heart rate, systolic, diastolic and mean arterial blood pressure will be recorded at same measuring points and during recruitment.

Assessment for incidence of pneumothorax and postoperative pulmonary complications like; postoperative lung collapse and postoperative pneumonia.

Assessment the duration of postoperative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II.
2. Age (1-4) years.
3. Patients undergoing major abdominal surgery in supine position (eg. Splenectomy, exploration, kasai etc.,).

Exclusion Criteria:

1. Parents' refusal.
2. Patients with congenital heart disease.
3. Patients with chronic pulmonary disease ( asthma, bronchiectasis, emphysematous disease, etc.,)
4. Patients with respiratory tract infection.
5. Patients with chest wall deformities

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
The lung aeration score 5minutes following induction of general anesthesia | Lung ultrasound examinations will be performed 5minutes following induction of general anesthesia
  Atelectasis will be assessed by ultrasound using lung aeration score applied for each region. Lung score is four points (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation) so, applying score for 12 regions bilateral will result in maximum score 36 and lowest score 0

SECONDARY OUTCOMES:
•The sum of surface area of atelectatic regions | It will be measured at different time-points immediately before induction of anesthesia, 5, 15 minutes following induction of general anesthesia,5 min before extubation and 5 min after extubation at recovery room to detect and monitor atelectasis
  The sum of surface area of atelectatic regions and the number of recruitment attempts to recruit atelectatic areas will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Iman R Abdel- Aal, Professor, Study Director — Anesthesia department , Cairo university
Locations (1):
- Kasr Alainy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No